CLINICAL TRIAL: NCT04304651
Title: Screening for Occult Malignancy Using 18F-Fluorodeoxyglucose Positron Emission Tomography/Computed Tomography (FDG PET/CT) in Patients with Unprovoked Venous Thromboembolism
Brief Title: Screening for Occult Malignancy in Patients with Unprovoked Venous Thromboembolism
Acronym: MVTEP2/SOME2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Ministry of Health, France (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government); Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 29BRC20.0021
Record Dates: First submitted 2020-03-07; First posted 2020-03-11 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Embolism and Thrombosis
Keywords: venous thrombosis; pulmonary embolism; screening; occult cancer
MeSH Terms: conditions — Embolism and Thrombosis; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Limited cancer screening (Active Comparator): Limited screening alone.
  Interventions: Diagnostic Test: Limited cancer screening
- Limited cancer screening + FDG PET/CT (Experimental): Limited screening + FDG PET/CT
  Interventions: Diagnostic Test: Limited cancer screening + FDG PET/CT

INTERVENTIONS:
Diagnostic Test: Limited cancer screening — The limited cancer screening will include: 1) a complete medical history and physical examination; 2) complete blood count; 3) liver function tests (AST, ALT, ALP, bilirubin); and 4) chest X-ray.
  In women, a breast examination, Pap smear/pelvic examination (if < 70 years old and previously sexually active) and mammogram will be performed, if not conducted in last year.
  In men, similarly, prostate examination and PSA testing will be performed, if not conducted in the last year.
  All patients will undergo colon cancer screening as per local practice.
  Arms: Limited cancer screening
Diagnostic Test: Limited cancer screening + FDG PET/CT — The limited cancer screening (as described above) in combination with a FDG PET/CT.
  Arms: Limited cancer screening + FDG PET/CT

SUMMARY:
Venous thromboembolism (VTE) can be the earliest sign of cancer. Identifying occult cancers at the time of VTE diagnosis may lead to significant improvement of patients' care. This is also an upmost issue for patients who want to know if an underlying cancer might have triggered the VTE.

An individual patient-level data meta-analysis (IPDMA) supports extensive screening strategies for occult cancer especially based on FDG PET/CT, and suggests that the best target population for cancer screening would be patients with unprovoked VTE older than 50 years of age (6.7% in patients aged 50 years or more vs. 1.0% in patients of less than 50 years (OR: 7.1, 95% CI: 3.1 to 16%).

DETAILED DESCRIPTION:
The identification of subgroups of patients at high risk of cancer might enable more efficient screening strategies for early detection of cancer. Venous thromboembolism (VTE) can be the first manifestation of an occult cancer. All tumor sites may be involved. In an individual patient-level data meta-analysis (IPDMA), it was reported a 1-year prevalence of occult cancer of 5.2% (95%CI 4.1-6.5) among patients presenting with unprovoked VTE.

Two recent multicenter randomized controlled trials (e.g. SOME (Canada) and MVTEP (France) trials) failed to demonstrate that extensive cancer screening strategies diagnosed more cancers, more early stage tumors, or improved cancer-related mortality in comparison with a more limited screening strategy. However, the main limitation of these studies was the twice lower than expected overall incidence of occult cancer diagnosis in unselected patients with unprovoked VTE, which limited the statistical power. In the IPDMA, it was also reported that the 1-year period prevalence of occult cancer was 7-fold higher in patients aged ≥ 50 (6.8%; 95%CI 5.6-8.3) as compared with those < 50 years (1.0%; 95%CI 0.5-2.3).

Moreover, in the MVTEP trial, the incidence of missed cancers over a 2-years follow-up period was significantly lower in patients randomized to a 18F-Fluorodeoxyglucose Positron Emission/Computed Tomography (FDG-PET/CT) screening strategy. Thus, the most promising diagnostic modality for occult cancer screening seems to be FDG-PET/CT. FDG-PET/CT which allows a one-stop whole-body imaging, is routinely used for the diagnosis, staging and restaging of various cancers.

The MVTEP2 Trial seeks to determine if among higher risk patients (≥ 50 year-old) with a first unprovoked VTE, a cancer screening strategy including a FDG-PET/CT decreases the number of missed occult cancers detected over a 1-year follow-up period as compared with a limited screening alone.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 50 years or older with a new diagnosis of first unprovoked proximal deep vein thrombosis (DVT) and/or pulmonary embolism (PE) will be eligible to participate into the study.

Unprovoked VTE is defined as the absence of any of the following predisposing factors:

1. active malignancy (known malignancy, progressive and/or treated during the last 5 years) except for adequately treated basal or squamous cell carcinoma; Patients whose state of health suggests the presence of cancer at the time of diagnosis of VTE cannot be included in the protocol
2. recent (less than 3 months) paralysis, paresis or plaster immobilization of the lower extremities;
3. recently bedridden for period of 3 or more days, or major surgery, within the previous 12 weeks requiring general or regional anaesthesia;
4. previous unprovoked VTE;
5. known thrombophilia (hereditary or acquired)

Exclusion Criteria:

Patients will be excluded from the study if they have any of the following criteria:

1. Refusal or inability to provide informed consent;
2. Hypersensitivity to 18F-FDG or any of the excipients according to the product monograph;
3. Unavailable to follow-up.
4. VTE while on anticoagulation (e.g apixaban, rivaroxaban, edoxaban, dabigatran, warfarin)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1276 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2026-09-08 (Estimated); Study Completion 2030-09-08 (Estimated)

PRIMARY OUTCOMES:
Occult cancer missed by screening strategies | At 1 year of follow-up
  Occult cancer "missed" by cancer screening defined as proven cancer diagnosed (either biopsy proven cancer or cancer diagnosis approved by adjudication committee in the absence of biopsy proven cancer) from the time of cancer screening completion to the end of the 1-year follow-up period, and not detected at the time of screening. In other words, "missed" means the number of new cancers diagnosed in patients considered not to have cancer after having completed the assigned cancer screening strategy (i.e false negative results of screening strategies).

SECONDARY OUTCOMES:
Occult cancer diagnosed by screening strategies | At 1 month
  The proportion of patients with a new cancer diagnosis after completion of the initial allocated screening strategy.
Early vs Adanced-stage cancers | At 1 year of follow-up
  The proportion of early-stage (T1-2N0M0) as per the World Health Organization TNM classification system) versus advanced-stage tumors at initial screening and during follow-up.
Cancer-related mortality | At 5 years of follow-up
  Cancer-related mortality during a 5-year follow-up period.
Cost effectiveness analysis | At 1 year of follow-up
  Additional cost per additional cancer detected.
Recurrent VTE | At 1 year of follow-up
  Rate of recurrent VTE
Decision aid to assist patients in the decision of cancer screening | At 1 year of follow-up
  Development of a decision aid to assist patients in the decision of cancer screening
Additional tests | At 1 year of follow-up
  The proportion of patients receiving additional tests following each strategy

CONTACTS AND LOCATIONS:
Locations (20):
- Canada (10):
  - University of Calgary, Calgary, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - McMaster University, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Hopital Montfort, Ottawa, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
- France (10):
  - CH des Pays de Morlaix, Morlaix, France
  - CH Agen, Agen
  - CHU Angers, Angers
  - Brest University Hospital, Brest
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - CHU de Limoges, Limoges
  - Hôpital Européen Georges Pompidou, Paris
  - CHU Saint-Etienne, Saint-Etienne
  - Hôpital Saint Musse - CH Toulon, Toulon

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Background] Robin P, Le Roux PY, Planquette B, Accassat S, Roy PM, Couturaud F, Ghazzar N, Prevot-Bitot N, Couturier O, Delluc A, Sanchez O, Tardy B, Le Gal G, Salaun PY; MVTEP study group. Limited screening with versus without (18)F-fluorodeoxyglucose PET/CT for occult malignancy in unprovoked venous thromboembolism: an open-label randomised controlled trial. Lancet Oncol. 2016 Feb;17(2):193-199. doi: 10.1016/S1470-2045(15)00480-5. Epub 2015 Dec 8. PMID 26672686
- [Background] Carrier M, Lazo-Langner A, Shivakumar S, Tagalakis V, Zarychanski R, Solymoss S, Routhier N, Douketis J, Danovitch K, Lee AY, Le Gal G, Wells PS, Corsi DJ, Ramsay T, Coyle D, Chagnon I, Kassam Z, Tao H, Rodger MA; SOME Investigators. Screening for Occult Cancer in Unprovoked Venous Thromboembolism. N Engl J Med. 2015 Aug 20;373(8):697-704. doi: 10.1056/NEJMoa1506623. Epub 2015 Jun 22. PMID 26095467
- [Background] van Es N, Le Gal G, Otten HM, Robin P, Piccioli A, Lecumberri R, Jara-Palomares L, Religa P, Rieu V, Rondina M, Beckers MM, Prandoni P, Salaun PY, Di Nisio M, Bossuyt PM, Buller HR, Carrier M. Screening for Occult Cancer in Patients With Unprovoked Venous Thromboembolism: A Systematic Review and Meta-analysis of Individual Patient Data. Ann Intern Med. 2017 Sep 19;167(6):410-417. doi: 10.7326/M17-0868. Epub 2017 Aug 22. PMID 28828492